CLINICAL TRIAL: NCT02170597
Title: Bioavailability of BIBR 953 ZW After 150 mg of BIBR 1048 (Oral Pro-drug of BIBR 953 ZW) Administered as HPMC Capsule Relative to a Gelatine Capsule, and Bioavailability of the HPMC Capsule Under the Influence of Food in Healthy Subjects. A Three-way Crossover, Randomised, Open Trial
Brief Title: Bioavailability of BIBR 953 ZW Under Influence of Food in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.40
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (3):
- BIBR 1018 MS HPMC capsule fasted (Experimental)
  Interventions: Drug: BIBR 1048 MS HPMC capsule
- BIBR 1048 MS HPMC capsule after high fat meal (Experimental)
  Interventions: Drug: BIBR 1048 MS HPMC capsule
- BIBR 1048 MS gelatine capsule fasted (Active Comparator)
  Interventions: Drug: BIBR 1048 MS gelatine capsule

INTERVENTIONS:
Drug: BIBR 1048 MS HPMC capsule
  Arms: BIBR 1018 MS HPMC capsule fasted; BIBR 1048 MS HPMC capsule after high fat meal
Drug: BIBR 1048 MS gelatine capsule
  Arms: BIBR 1048 MS gelatine capsule fasted

SUMMARY:
Study to investigate the relative bioavailability of BIBR 953 ZW after administration of a 150 mg BIBR 1048 HPMC (hydroxypropylmethylcellulose) capsule versus BIBR 953 ZW after administration of a 150 mg BIBR 1048 gelatine capsule, and to investigate the relative bioavailability of BIBR 953 ZW given as BIBR 1048 MS HPMC capsule with food versus without food.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with GCP and local legislation
* Age ≥ 18 and ≤ 55 years
* BMI ≥ 18.5 and ≤ 29.9 kg/m2

Exclusion Criteria:

* Any finding at the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History of or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of relevant orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of:

  * allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * any bleeding disorder including prolonged or habitual bleeding
  * other hematologic disease
  * cerebral bleeding (e.g. after a car accident)
  * commotio cerebri
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs that might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* History of any familial bleeding disorder
* Thrombocytes < 150000/μl

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2003-08; Primary Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the plasma concentration time curve from zero time extrapolated to infinity) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug
AUC0-tz (The area under the plasma concentration time curve from zero time to the time of the last quantifiable concentration) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug
Cmax (maximum measured concentration) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug
tmax (time from dosing to when the plasma concentration reaches Cmax after extravascular doses) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug

SECONDARY OUTCOMES:
t½ (terminal half-life) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug
MRT (Total mean residence time) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug
CL/F (Total apparent clearance) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug
Vz/F (Apparent volume of distribution) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug